CLINICAL TRIAL: NCT03254745
Title: Evaluation of Pharmacist's Intervention in Improving Treatment Outcomes of Rheumatoid Arthritis Patients in Karachi, Pakistan: The Pharmacist Assisted Care Trial for Rheumatoid Arthritis Patients (PACTRA)
Brief Title: Evaluation of Pharmacist's Intervention in Improving Treatment Outcomes of Rheumatoid Arthritis: A Randomized Controlled Trial
Acronym: PACTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Atta Abbas Naqvi, Atta Abbas Naqvi, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PACT1
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Pakistan; Pharmacist; Intervention; Treatment outcome
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator will be blinded. Outcome assessor would be blinded. Patients in the control group would be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist intervention (Experimental): 1. Disease education (General education about rheumatoid arthritis in a verbal and written manner)
  2. Dietary and lifestyle modifications (General recommendations as well as specific ones based on patients' baseline health status)
  3. Counseling regarding adherence (General lecture on adherence to medications and physical rehabilitation in rheumatoid arthritis as well as specific advice based on patients health status)
  4. Advice on medication use (General counseling on medication use as well as patient centered counseling).
  Interventions: Other: Pharmacist led pharmaceutical care
- Usual care (No Intervention): Patients will not be counseled by pharmacist and will be allowed to take usual care.

INTERVENTIONS:
Other: Pharmacist led pharmaceutical care — The intervention in the study will be a pharmacist's intervention that will be provided to rheumatoid arthritis patients in order to improve their treatment outcomes. It will be in the form of a single (1) session by pharmacist (face-to-face) followed by written material for use at home. The pharmacist will look at the patient's baseline data and provide counseling. The venue for counseling will be the hospitals.
  Arms: Pharmacist intervention

SUMMARY:
Rheumatoid arthritis is an auto-immune disorders that mainly affects the joints. It may also affect other organs of the body such as skin, eyes, lungs and heart. The immune system of the body attacks the lining of the joint that results in erosion and joint deformity. This condition if untreated may lead to disability. RA is managed by medications known as disease modifying anti rheumatic drugs (DMARDs) as well as physical therapy. Dietary and lifestyle modification may also ease the condition.

DETAILED DESCRIPTION:
One of the major problems in managing RA is adherence to rehabilitation and medication. Studies report low adherence to medication among patients of RA. Certain barriers to rehabilitation also exists which may include exhaustive treatment attendance, time management and direct costs. Patient intentionally make decisions of non adherence to their prescribed rehabilitation schedule and medication regimen. This may be due to suffering from adverse drug reactions (ADRs) of medications, excessive pain arising from physical therapy and/or out-of-pocket costs.

Pharmacists have the potential to improve the patient's clinical, humanistic and economic outcomes in rheumatoid arthritis by providing pharmaceutical care. This can be executed by:

1. Resolving drug related problems and managing drug therapy
2. Management of modifiable risk factors such as weight
3. Recommending dietary and lifestyle changes
4. Providing patient counseling, disease education and medication advice
5. Reducing the out-of-pocket costs
6. Improve overall well being and quality of life

Evidence from the past indicates a varying prevalence of RA in Pakistan. Figures for prevalence of RA varied geographically as literature reported a prevalence of 0.142% to 5.5% in the southern and northern region of Pakistan respectively. Recently, a study conducted in a tertiary care unit in the city of Karachi located in southern region reported a figure of 633 (12.9%) for RA patients out of total 4900 patients who visited rheumatology clinic in the hospital. It highlighted that disease burden in this region has dramatically increased.

Most Pakistani patients lack adequate disease knowledge and awareness regarding RA. Moreover, patients in Pakistan have to pay direct medical cost in most of the cases. In the past, studies have highlighted that Pakistani patients view costs per session and treatment attendance as major barriers to undergo physical therapy sessions for rheumatological disorders.

There is a dearth of literature reported on pharmacist's inclusion to improve treatment outcomes in rheumatoid arthritis.There are no reported figures for adherence to treatment and medications for RA or any musculoskeletal disease. Studies conducted in Pakistan also highlight that pharmacists have the potential to improve economic, clinical and humanistic outcomes by providing pharmaceutical care to patients. However, it is to be seen if pharmacist can actually achieve the milestone i.e. improve patient treatment outcomes of rheumatoid arthritis. A randomized trial is therefore needed employing pharmacist intervention in RA patients. This present an excellent opportunity to identify the areas where a pharmacist has the potential to play his/her role and evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients with established diagnosis of rheumatoid arthritis over 3 months.
* Participants who are willing to participate in the study.

Exclusion Criteria:

* Patients with no rheumatoid arthritis.
* Patients currently undergoing surgery or had previous history of surgery.
* Patients with more than 3 comorbidities.
* Patients who are not willing to participate.
* In-patients will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Disease knowledge | Week 12 from baseline
  Knowledge about rheumatoid arthritis
Medication Adherence | Week 12 from baseline
  Patients' adherence to their medications
Health Related Quality of Life (HR-QOL) | Week 12 from baseline
  Rheumatoid arthritis patients' health related quality of life
Treatment Adherence | Week 12 from baseline
  Patients' adherence to their rehabilitation
Direct Cost of treatment | Week 12 from baseline
  Direct cost of rheumatoid arthritis treatment on patient's pocket
Disease Activity | Week 12 from baseline
  The disease activity was assessed by disease activity score (DAS) also known as DAS - 28 score.
Adverse events | Week 12 from baseline
  The adverse events were assessed directly through patients' medical history that was available in hospital database.

SECONDARY OUTCOMES:
Patient satisfaction | At Week 12
  Patient satisfaction from pharmacists in managing rheumatoid arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Azmi A Hassali, PhD, Study Director — Universiti Sains Malaysia
Locations (1):
- Clifton Central Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No